CLINICAL TRIAL: NCT07053436
Title: MMRC Horizon Two: A Phase II Randomized Adaptive Platform Trial Integrating Novel Therapies in High-Risk-Newly Diagnosed Multiple Myeloma
Brief Title: Horizon Two Adaptive Platform Study in High Risk Newly Diagnosed Multiple Myeloma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Multiple Myeloma Research Consortium (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMRC-100
Record Dates: First submitted 2025-05-28; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: High Risk Newly Diagnosed Multiple Myeloma
Keywords: Horizon; Horizon Two; MMRC; HR NDMM
MeSH Terms: interventions — Antibodies, Bispecific; Antibodies, Monoclonal; Stem Cell Transplantation; isatuximab

STUDY DESIGN:
Intervention Model Description: Adaptive Platform
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control Arm: Isa-KRd with Autologous Stem Cell Transplant (Active Comparator): Appendix A to the MMRC Horizon Two High Risk Newly Diagnosed Multiple Myeloma Master Protocol: Isa-KRd with Autologous Stem Cell Transplant in Patients with High Risk Newly Diagnosed Multiple Myeloma
  Interventions: Drug: Monoclonal Antibody with Stem Cell Transplant
- Induction, Consolidation, and Maintenance Therapy Combining Linvoseltamab and Triplet Therapy (Experimental): Appendix B to the MMRC Horizon Two High Risk Newly Diagnosed Multiple Myeloma Master Protocol: Induction, Consolidation, and Maintenance Therapy Combining Linvoseltamab and Triplet Therapy in Patients with High Risk Newly Diagnosed Multiple Myeloma
  Interventions: Drug: Bispecific Monoclonal Antibody and Triplet Therapy

INTERVENTIONS:
Drug: Bispecific Monoclonal Antibody and Triplet Therapy — Induction, Consolidation, and Maintenance Therapy Combining Linvoseltamab and Triplet Therapy
  Other Names: Linvoseltamab
  Arms: Induction, Consolidation, and Maintenance Therapy Combining Linvoseltamab and Triplet Therapy
Drug: Monoclonal Antibody with Stem Cell Transplant — Isatuximab-KRd with Autologous Stem Cell Transplant
  Other Names: Isatuximab
  Arms: Control Arm: Isa-KRd with Autologous Stem Cell Transplant

SUMMARY:
The Multiple Myeloma Research Consortium (MMRC) Horizon Two trial is a master protocol, multi-center, phase II randomized adaptive platform trial designed to efficiently evaluate multiple investigational therapies in high-risk newly diagnosed multiple myeloma patients using an integrated and patient-centric clinical research platform that enables longitudinal learning and sharing of knowledge and investigates multiple novel therapeutic strategies within one trial platform.

DETAILED DESCRIPTION:
The master protocol has broad scope and substantial flexibility, allowing each investigational arm within the platform to have its own design. The master protocol specifies general principles but the analysis plan for each investigational arm will be specified in its appendix. Details outlined in each investigational arm's appendix will include any co-primary endpoints (if applicable), the comparator arm, sample size and justification, inclusion of a safety run-in (if required), and any potential adaptations within the appendix. Accrual to an investigational arm will terminate in accord with its appendix.

As an adaptive platform trial, MMRC Horizon Two will evaluate multiple investigational arms against common controls. It is expected that the common controls may vary over time as standard of care therapy evolves. An initial common control arm will be specified in the control arm appendix. Changes in the common controls will be made through amendments to this appendix.

All patients will be randomized to an arm in the study. The default for the platform will be equal randomization to all arms that a patient is eligible. However, when there are more than two investigational arms and response adaptive randomization is deemed beneficial, it may be implemented in the trial.

Participants will be on study for 5 years from the date of randomization, inclusive of treatment and follow-up periods. Specifics on treatment duration and duration of follow up will be included in the respective arm appendix.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agree to participate by giving written informed consent

  -≥18 years of age
* Symptomatic and transplant eligible newly diagnosed multiple myeloma histologically confirmed per IMWG criteria that is high-risk as defined by at least one of the following:

  * Del(17p) (CCF ≥ 20%, by analyses conducted on CD138-positive/purified cells) and/or TP53 mutation assessed by NGS
  * One of these translocations-t(4;14) or t(14;16) or t(14;20)-co-occurring with +1q and/or del(1p32)
  * Monoallelic del(1p32) along with +1q, or biallelic del(1p32)
  * High β2M (≥5.5 mg/dL) with normal creatinine (<1.2 mg/dL)
  * Presence of extra-medullary disease non-contiguous with bone at diagnosis (by PET-CT or Whole Body MRI)
  * Primary plasma cell leukemia (circulating plasma cells > 5% at diagnosis)
* No more than 2 cycles of NCCN listed induction therapy for multiple myeloma
* Measurable disease, per IMWG criteria, at time of diagnosis defined as one of the following:

  * Serum M-protein at diagnosis ≥ 0.5g/dL (0.3 g/dL or above if IgA subtype)
  * Urine M-protein ≥ 200 mg/24hours
  * Serum free light chain difference > 100 mg/L
  * Plasmacytoma ≥ 2cm
  * Bone marrow involvement ≥ 30%
* ECOG performance status of 0-2
* Adequate organ function, as indicated by the following laboratory values:

  * Adequate hematological function, defined as ANC ≥ 1000/µL, platelet count ≥ 75,000/µL, and hemoglobin ≥ 8 g/dL (transfusion and/or growth factor support is allowed for hematologic parameters as long as the investigator deems the patient otherwise fit for screening)
  * Adequate hepatic function, defined as total bilirubin level ≤ 1.5 x institutional upper limit of normal (IULN) except in participants with congenital bilirubinemia, such as Gilbert syndrome (in which case direct bilirubin ≤1.5 x IULN is required), AST ≤ 2.5 x IULN, and ALT ≤ 2.5 x IULN
  * Adequate renal function, defined as calculated creatinine clearance ≥ 30 mL/min per institutional standard (assessment method should be recorded, measured or C-G acceptable)
* Persons of childbearing potential must have a negative serum pregnancy test at screening (within 72 hours of first dose of trial medication). Non-childbearing potential for a person assigned as female at birth is defined as 1 of the following:

  --≥ 45 years of age and has not had menses for >1 year
  * Amenorrheic for > 2 years without a hysterectomy and/or oophorectomy and follicle-stimulating hormone value in the postmenopausal range upon pretrial (screening) evaluation
  * Status is post-hysterectomy, -oophorectomy, or -tubal ligation
* Persons of childbearing potential must be willing to use highly effective contraceptive measures during sexual contact with a person assigned as male at birth starting with the Screening visit through 90 days after last dose of trial medication.

  --Note: Abstinence is acceptable if this is the established and preferred contraception for the participant.
* Persons assigned as male at birth with a partner(s) of childbearing potential must agree to use highly effective contraceptive measures throughout the trial starting with the Screening visit through 90 days after the last dose of trial medication is received. Persons assigned as male at birth with pregnant partners must agree to use a condom; no additional method of contraception is required for the pregnant partner.

  --Note: Abstinence is acceptable if this is the established and preferred contraception method for the participant.
* Known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using New York Heart Association Functional Classification. To be eligible for this trial, participants should be Class 2 or better. Class 2 is defined as slight limitation of physical activity, in which ordinary physical activity leads to fatigue, palpitation, or dyspnea; the person is comfortable at rest.
* Prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessments of the investigational arms are eligible for this trial.
* Known HIV infection and on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* Evidence of chronic hepatitis B virus (HBV) infection must have an undetectable HBV viral load on suppressive therapy, if indicated.
* History of hepatitis C virus (HCV) infection must have been treated and cured. For patients with known HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Willing and able to comply with the requirements of the protocol.

Exclusion Criteria:

* Major concurrent illness or organ dysfunction including but not limited to the following:

  * POEMS syndrome
  * Symptomatic major organ involvement AL amyloidosis
* History of allergy or known hypersensitivity to any of the trial therapies or any of their excipients, or contraindication to any of the trial therapies as outlined in the local prescribing information (e.g., United States Prescribing Information [USPI])
* Complete spinal cord compression or CNS involvement
* Known leptomeningeal disease
* Allogeneic tissue/solid organ transplant recipients with chronic GVHD requiring steroid equivalent dose of > 20 mg prednisone
* Active infection requiring treatment
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or is not in the best interest of the participant to participate, in the opinion of the treating investigator
* Psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the trial
* Legally incapacitated or has limited legal capacity
* Persons who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2035-10-01 (Estimated); Study Completion 2035-10-12 (Estimated)

PRIMARY OUTCOMES:
Sustained measurable residual disease (MRD) negativity | 2 years post randomization
  Sustained MRD negativity is defined as MRD negativity at a minimum threshold of one myeloma cell in one hundred thousand nucleated bone marrow cells at MRD assessments
Progression Free Survival | through study completion, roughly 5 years
  PFS is defined as time from randomization to disease progression or death from any cause. Participants who have not progressed or died are censored at the date last known progression-free.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 2 years
  ORR is defined as the percentage of people who have achieved a partial response (PR) or better according to the IMWG criteria within the defined period of time on trial.
Best overall response | 2 years
  Best overall response (Stringent Complete Response [sCR], Complete Response [CR], Very Good Partial Response [VGPR], Partial Response [PR], Stable Disease [SD], Progressive Disease [PD]) by International Myeloma Working Group Response Criteria.
Two-year progression free survival rate | 24 months after randomization
  Two-year progression free survival rate is defined as the proportion of participants alive and progression-free 24 months after randomization.
Overall survival (OS) | through study completion, average of 5 years
  OS is defined as the time from randomization to death. Alive participants are censored at the date last known alive.
Duration of response (DoR) | 2 years
  DoR is defined as time from the first observation of a confirmed response [Stringent Complete Response (sCR), Complete Response (CR), Very Good Partial Response (VGPR), or Partial Response (PR)] to first documentation of disease progression or death. Participants who have not progressed or died are censored at the date last known progression-free. The start date for DoR is the date the response was first observed, not the date of confirmation.
12-month measurable residual disease (MRD) negativity | 12 months from randomization
  12-month MRD negativity is defined as MRD negativity at a minimum threshold of one myeloma cell in one hundred thousand nucleated bone marrow cells at MRD assessment at disease restaging 1 (12 months±3 months from randomization). Measured using ClonoSEQ's standardized, commercial, next generation sequencing assay (preferred) or commercial multi-color flow cytometry.
Frequency and intensity of (serious) adverse events (S)AEs | through study completion, an average of 5 years
  Assessed by NCI CTCAE version 5.0, including a focus on hematologic clinical laboratory abnormalities and changes.

CONTACTS AND LOCATIONS:
Overall Officials: Hearn Jay Cho, MD, PhD, Principal Investigator — Multiple Myeloma Research Foundation

IPD SHARING:
Plan to Share IPD: Undecided